CLINICAL TRIAL: NCT02287844
Title: Xylo-oligosaccharide (XOS) in Combination With Inulin Modulates Both the Intestinal Environment and Immune Status in Healthy Subjects, While XOS Alone Only Shows Prebiotic Properties
Brief Title: Prebiotics Change Microflora and Decrease LPS
Acronym: PIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: Institut Polytechnique LaSalle Beauvais (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, MD, Nutritionist, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2007-A00273-50
Record Dates: First submitted 2014-11-04; First posted 2014-11-11 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Prebiotics Effect
Keywords: Xylo-oligosaccharides; Immunonutrition; Prebiotics; Lipopolysaccharides; Cytokines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- XOS group (Experimental): Subjects consumed 6.64 g of a XOS-enriched compound derived from wheat arabinoxylans (5 g of XOS) everyday for 4 weeks.
  Interventions: Other: XOS
- INU-XOS group (Experimental): Subjects consumed 6.64 g of a mixture containing inulin-type fructans, XOS and maltodextrins (3 g of inulin and 1 g of XOS) everyday for 4 weeks.
  Interventions: Other: INU-XOS
- Placebo (Active Comparator): Subjects consumed 6.64 g of wheat maltodextrins everyday for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: XOS — 5 g of XOS everyday for 4 weeks.
  Arms: XOS group
Other: INU-XOS — 1 g of XOS and 3 g of inulin everyday for 4 weeks.
  Arms: INU-XOS group
Other: Placebo — 6.64 g of maltodextrins everyday for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of the present study was to establish the prebiotic effect of a new xylo-oligosaccharides (XOS) and of an inulin-and-XOS mixture (INU-XOS) and to determine their effect on endotoxaemia (lipopolysaccharides (LPS)) and immune parameters. In this randomized, parallel, placebo-controlled, double-blind study, sixty healthy volunteers were randomly assigned to three groups, receiving either 5 g XOS, INU-XOS (3 g inulin +1 g XOS) or an equivalent weight of wheat maltodextrins (placebo) during 4 weeks.

DETAILED DESCRIPTION:
The study followed a randomized, parallel placebo-controlled double-blind design.

A semi-quantitative dietary survey was performed at enrollment in order to assess the usual dietary fiber intake in order to select the target population consuming 13 to 18 g/day. The volunteers were instructed to follow dietary guidelines to maintain their fiber intake during a two-week stabilization phase and then throughout the intervention.

As all volunteers were living on-site and taking all meals at the Institut Polytechnique LaSalle Beauvais cafeteria, the content of each meal could be closely controlled during the week. A 3-day dietary survey was performed at the end of the stabilization period and repeated at the end of the intervention in order to assess the stability of the diet.

The 60 volunteers were randomly assigned to one of three groups and received daily the intervention for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Stable weight (+/- 3 kg) for the last 3 months
* Body Mass Index (BMI) between 18.5 and 27 kg/m²
* Consuming between 13 and 18 g of dietary fiber a day
* Student on campus at the Institut Polytechnique LaSalle Beauvais
* Informed consent form signed
* Able to follow the requirement of the study
* Have a social security

Exclusion Criteria:

* Has a serious pathology
* Has a gastrointestinal, vesicular or pancreatic disease
* Took an antibiotic or a laxative treatment in the last 6 months
* Surgery of the gastrointestinal tract in the last 12 months
* Orange juice intolerance
* Chronic or recurring diarrhea, constipation or abdominal pain
* Taking drugs known to have an effect on the gastrointestinal, pancreatic and vesicular function
* Recent gastroenteritis or foodborne illness
* Diabetes
* Consuming regularly of probiotics- or prebiotics-enriched products in the last month
* Drinking more than 3 glasses of alcohol a day
* Is deprived of liberty
* Is under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the intestinal bifidobacterium at 4 weeks. | 4 weeks
  Dosage by count in the feces by Reverse transcription polymerase chain reaction (RT-PCR).

SECONDARY OUTCOMES:
Change from Baseline in the intestinal bifidobacterium at 2 weeks. | 2 weeks
  Dosage by count in the feces by Reverse transcription polymerase chain reaction (RT-PCR).
Change from 2 weeks in the intestinal bifidobacterium at 4 weeks. | Between 2 and 4 weeks
  Dosage by count in the feces by Reverse transcription polymerase chain reaction (RT-PCR).
Change from Baseline in total microbiota and composition in the feces at 4 weeks. | 4 weeks
  Total bacterial count and specific bacterial profile analyzed by quantitative PCR.
Change from Baseline in total microbiota and composition in the feces at 2 weeks. | 2 weeks
  Total bacterial count and specific bacterial profile analyzed by quantitative PCR.
Change from 2 weeks in total microbiota and composition in the feces at 4 weeks. | Between 2 and 4 weeks
  Total bacterial count and specific bacterial profile analyzed by quantitative PCR.
Change from Baseline of short-chain fatty acids (C2, C3, C4) in the feces at 4 weeks | 4 weeks
  Acetic acid (C2), propionic acid (C3) and butyric acid (C4) extracted and measured.
Change from Baseline of short-chain fatty acids (C2, C3, C4) in the feces at 2 weeks | 2 weeks
  Acetic acid (C2), propionic acid (C3) and butyric acid (C4) extracted and measured.
Change from 2 weeks of short-chain fatty acids (C2, C3, C4) in the feces at 4 weeks | Between 2 and 4 weeks
  Acetic acid (C2), propionic acid (C3) and butyric acid (C4) extracted and measured.
Change from Baseline in the alpha-glucosidase and beta-glucuronidase activities in the feces at 4 weeks. | 4 weeks
Change from Baseline in the alpha-glucosidase and beta-glucuronidase activities in the feces at 2 weeks. | 2 weeks
Change from 2 weeks in the alpha-glucosidase and beta-glucuronidase activities in the feces at 4 weeks. | Between 2 and 4 weeks
Change from Baseline in the phenol and p-Cresol in the feces at 4 weeks. | 4 weeks
Change from Baseline in the phenol and p-Cresol in the feces at 2 weeks. | 2 weeks
Change from 2 weeks in the phenol and p-Cresol in the feces at 4 weeks. | Between 2 and 4 weeks
Change from Baseline in the faecal pH and dry matter at 4 weeks. | 4 weeks
Change from Baseline in the faecal pH and dry matter at 2 weeks. | 2 weeks
Change from 2 weeks in the faecal pH and dry matter at 4 weeks. | Between 2 and 4 weeks
Change from Baseline in secretory Immunoglobulin A (IgA) at 4 weeks. | 4 weeks
  Measured with s-IgA ELISA kit.
Change from Baseline in secretory Immunoglobulin A (IgA) at 2 weeks. | 2 weeks
  Measured with s-IgA ELISA kit.
Change from 2 weeks in secretory Immunoglobulin A (IgA) at 4 weeks. | Between 2 and 4 weeks
  Measured with s-IgA ELISA kit.
Change from Baseline in cytokines at 4 weeks | 4 weeks
  Tumor Necrosis Factor (TNF)-alpha and Interleukine(IL)-10
Change from Baseline in cytokines at 2 weeks | 2 weeks
  Tumor Necrosis Factor (TNF)-alpha and Interleukine(IL)-10
Change from 2 weeks in cytokines at 4 weeks | Between 2 and 4 weeks
  Tumor Necrosis Factor (TNF)-alpha and Interleukine(IL)-10
Change from Baseline in dietary intakes at 4 weeks | 4 weeks
  Data extracted from a 3-day food diary.
Change from Baseline in dietary intakes at 2 weeks | 2 weeks
  Data extracted from a 3-day food diary.
Change from 2 weeks in dietary intakes at 4 weeks | Between 2 and 4 weeks
  Data extracted from a 3-day food diary.
Change from Baseline of circulating lipopolysaccharides (LPS) at 4 weeks. | 4 weeks
  Measured in plasma sample using the limulus amebocyle lysate chromogenic endpoint assay.
Change from Baseline of circulating lipopolysaccharides (LPS) at 2 weeks. | 2 weeks
  Measured in plasma sample using the limulus amebocyle lysate chromogenic endpoint assay.
Change from 2 weeks of circulating lipopolysaccharides (LPS) at 4 weeks. | Between 2 and 4 weeks
  Measured in plasma sample using the limulus amebocyle lysate chromogenic endpoint assay.
Change from Baseline in the subjects' tolerance to the test products at 4 weeks. | 4 weeks
  Flatulence, bloating, rumbling, cramps, nausea, stool consistency on a Visual Analog Scale (10 cm).Stool frequency (stool per day).
Change from Baseline in the subjects' tolerance to the test products at 2 weeks. | 2 weeks
  Flatulence, bloating, rumbling, cramps, nausea, stool consistency on a Visual Analog Scale (10 cm). Stool frequency (stool per day).
Change from 2 weeks in the subjects' tolerance to the test products at 4 weeks. | Between 2 and 4 weeks
  Flatulence, bloating, rumbling, cramps, nausea, stool consistency on a Visual Analog Scale (10 cm). Stool frequency (stool per day).

OTHER OUTCOMES:
Change from Selection (at least 2 weeks before Baseline) in Weight, Height, BMI, Blood pressure, Heart rate at 4 weeks | 4weeks
Change from Selection (at least 2 weeks before Baseline) in Weight, Height, BMI, Blood pressure, Heart rate at 2 weeks | 2 weeks
Change from 2 weeks in Weight, Height, BMI, Blood pressure, Heart rate at 4 weeks | Between 2 and 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Polytechnique LaSalle Beauvais, Beauvais, Oise, France